CLINICAL TRIAL: NCT02960776
Title: Effect of Long Term Sleep Restriction on Energy Balance
Brief Title: Impact of Sleep Restriction on Performance in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: NYU Langone Health (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Marie-Pierre St-Onge, Associate Professor of Nutritional Medicine, Columbia University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: AAAQ7746; 1R01HL128226-01A1 (NIH)
Record Dates: First submitted 2016-11-07; First posted 2016-11-10 (Estimated); Results first posted 2024-07-09 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Sleep; Obesity; Sleep Restriction
Keywords: Body Weight; Habitual sleep
MeSH Terms: conditions — Obesity; Body Weight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Habitual Sleep (HS) (No Intervention): Participants will be asked to follow a fixed bedtime routine based on the participant's regular bed- and wake-times during the habitual sleep (HS) phase.
- Sleep Restriction (SR) (Experimental): Participants will be asked to keep their habitual wake time constant but delay their bedtime to achieve a reduction of 1.5 hours in total sleep time during the sleep restriction (SR) phase.
  Interventions: Behavioral: Sleep Restriction (SR)

INTERVENTIONS:
Behavioral: Sleep Restriction (SR) — Participants will be asked to keep their habitual wake time constant but delay their bedtime to achieve a reduction of 1.5 hours in total sleep time. A delay in bedtimes was chosen rather than advancing wake-up time because it most closely reflects differences in sleep timing behavior between short and normal sleepers.
  Arms: Sleep Restriction (SR)

SUMMARY:
The overall goal of this project is to look at the effects of long-term, sustained sleep restriction (SR) in adults, and assess the effects on mood and cognitive and physical performance.

DETAILED DESCRIPTION:
Chronic Sleep Restriction (SR) is highly prevalent in today's modern society. Artificial light, portable electronic devices, and 24-h services have allowed individuals to remain active throughout the night, leading to reductions in sleep duration. SSD has been linked to obesity and our laboratory has been interested in establishing whether sleep could be a causal factor in the etiology of obesity. Given the increasing prevalence of obesity over the past 5 decades, coinciding with the marked reduction in sleep duration, further exploration into the role of sleep as a risk factor for obesity could provide additional ammunition in the fight to prevent further increases in the incidence of obesity.

This study will be a randomized, crossover, outpatient SR study with 2 phases of 6 weeks each, with a 6 week wash-out period between the phases. Sleep duration in each phase will be the participant's regular bed- and wake times during the habitual sleep (HS) phase and HS minus 1.5 hours in the SR phase. During the HS phase, participants will be asked to follow a fixed bedtime routine based on their screening sleep schedule. During the SR phase, participants will be asked to keep their habitual wake time constant but delay their bedtime to achieve a reduction of 1.5 hours in total sleep time.

ELIGIBILITY:
Inclusion Criteria:

* BMI 25-29.9 kg/m2
* Have at least one obese parent
* Habitually sleep 7-9 hours a night
* Free of any current and past sleep and psychiatric disorders, including eating disorders, diabetes or Cardiovascular disease (CVD) (i.e., normal scores on: Pittsburgh Quality of Sleep Questionnaire Epworth Sleepiness Scale, Berlin Questionnaire, Sleep Disorders Inventory Questionnaire, Beck Depression Inventory, Composite Scale of Morningness/Eveningness, Three Factor Eating Questionnaire)
* All racial/ethnic groups

Exclusion Criteria:

* Smokers (any cigarettes or ex-smoker < 3 years)
* Neurological, medical or psychiatric disorder
* Diabetics
* Eating and/or sleep disorders
* Contraindications for MRI scanning
* Travel across time zones within 4 weeks
* History of drug and alcohol abuse
* Shift worker (or rotating shift worker)
* Caffeine intake > 300 mg/d
* Heavy equipment operators
* Commercial long-distance drivers

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2023-07-05 (Actual); Study Completion 2023-07-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Pierre St-Onge, PhD, Principal Investigator — Columbia University
Locations (1):
- New York Nutrition Obesity Research Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be provided on request after discussion among parties.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After study completion and publication of main findings.
Access Criteria: Contact PI for information

REFERENCES:
- [Background] Luckhaupt SE, Tak S, Calvert GM. The prevalence of short sleep duration by industry and occupation in the National Health Interview Survey. Sleep. 2010 Feb;33(2):149-59. doi: 10.1093/sleep/33.2.149. PMID 20175398
- [Background] Keith SW, Redden DT, Katzmarzyk PT, Boggiano MM, Hanlon EC, Benca RM, Ruden D, Pietrobelli A, Barger JL, Fontaine KR, Wang C, Aronne LJ, Wright SM, Baskin M, Dhurandhar NV, Lijoi MC, Grilo CM, DeLuca M, Westfall AO, Allison DB. Putative contributors to the secular increase in obesity: exploring the roads less traveled. Int J Obes (Lond). 2006 Nov;30(11):1585-94. doi: 10.1038/sj.ijo.0803326. Epub 2006 Jun 27. PMID 16801930
- [Background] Zuraikat FM, Makarem N, Redline S, Aggarwal B, Jelic S, St-Onge MP. Sleep Regularity and Cardiometabolic Heath: Is Variability in Sleep Patterns a Risk Factor for Excess Adiposity and Glycemic Dysregulation? Curr Diab Rep. 2020 Jul 23;20(8):38. doi: 10.1007/s11892-020-01324-w. PMID 32700156
- [Background] Makarem N, Zuraikat FM, Aggarwal B, Jelic S, St-Onge MP. Variability in Sleep Patterns: an Emerging Risk Factor for Hypertension. Curr Hypertens Rep. 2020 Feb 21;22(2):19. doi: 10.1007/s11906-020-1025-9. PMID 32086595
- [Result] Smith I, Salazar I, RoyChoudhury A, St-Onge MP. Sleep restriction and testosterone concentrations in young healthy males: randomized controlled studies of acute and chronic short sleep. Sleep Health. 2019 Dec;5(6):580-586. doi: 10.1016/j.sleh.2019.07.003. Epub 2019 Aug 12. PMID 31416797
- [Result] St-Onge MP, Campbell A, Salazar I, Pizinger T, Liao M, Aggarwal B. Information on Bedtimes and Wake Times Improves the Relation Between Self-Reported and Objective Assessments of Sleep in Adults. J Clin Sleep Med. 2019 Jul 15;15(7):1031-1036. doi: 10.5664/jcsm.7888. PMID 31383241
- [Result] Barragan R, Zuraikat FM, Tam V, Scaccia S, Cochran J, Li S, Cheng B, St-Onge MP. Actigraphy-Derived Sleep Is Associated with Eating Behavior Characteristics. Nutrients. 2021 Mar 5;13(3):852. doi: 10.3390/nu13030852. PMID 33807690
- [Result] Benasi G, Cheng B, Aggarwal B, St-Onge MP. The effects of sustained mild sleep restriction on stress and distress among healthy adults: Findings from two randomized crossover studies. Sleep Med. 2024 Mar;115:83-87. doi: 10.1016/j.sleep.2024.02.001. Epub 2024 Feb 2. PMID 38342031
- [Result] Zimmerman ME, Benasi G, Hale C, Yeung LK, Cochran J, Brickman AM, St-Onge MP. The effects of insufficient sleep and adequate sleep on cognitive function in healthy adults. Sleep Health. 2024 Apr;10(2):229-236. doi: 10.1016/j.sleh.2023.11.011. Epub 2024 Jan 16. PMID 38233280
- [Result] Li XY, Yoncheva Y, Yan CG, Castellanos FX, St-Onge MP. Chronic Mild Sleep Restriction Does Not Lead to Marked Neuronal Alterations Compared With Maintained Adequate Sleep in Adults. J Nutr. 2024 Feb;154(2):446-454. doi: 10.1016/j.tjnut.2023.12.016. Epub 2023 Dec 16. PMID 38104943
- [Result] Barragan R, Zuraikat FM, Cheng B, Scaccia SE, Cochran J, Aggarwal B, Jelic S, St-Onge MP. Paradoxical Effects of Prolonged Insufficient Sleep on Lipid Profile: A Pooled Analysis of 2 Randomized Trials. J Am Heart Assoc. 2023 Oct 17;12(20):e032078. doi: 10.1161/JAHA.123.032078. Epub 2023 Oct 10. PMID 37815115
- [Result] Barragan R, Zuraikat FM, Tam V, RoyChoudhury A, St-Onge MP. Changes in eating patterns in response to chronic insufficient sleep and their associations with diet quality: a randomized trial. J Clin Sleep Med. 2023 Nov 1;19(11):1867-1875. doi: 10.5664/jcsm.10696. PMID 37409467
- [Result] McAlpine CS, Kiss MG, Zuraikat FM, Cheek D, Schiroli G, Amatullah H, Huynh P, Bhatti MZ, Wong LP, Yates AG, Poller WC, Mindur JE, Chan CT, Janssen H, Downey J, Singh S, Sadreyev RI, Nahrendorf M, Jeffrey KL, Scadden DT, Naxerova K, St-Onge MP, Swirski FK. Sleep exerts lasting effects on hematopoietic stem cell function and diversity. J Exp Med. 2022 Nov 7;219(11):e20220081. doi: 10.1084/jem.20220081. Epub 2022 Sep 21. PMID 36129517
- [Derived] Petrov ME, Zuraikat FM, Cheng B, Aggarwal B, Jelic S, Laferrere B, St-Onge MP. Impact of sleep restriction on biomarkers of thyroid function: Two pooled randomized trials. Sleep Med. 2024 Dec;124:606-612. doi: 10.1016/j.sleep.2024.10.035. Epub 2024 Oct 30. PMID 39488926

RESULTS

PARTICIPANT FLOW:
Groups:
- Adequate Sleep Followed by Sleep Restriction: Participants were randomized to continue adequate sleep in phase 1 and crossed over to sleep restriction condition in phase 2
- Sleep Restriction Followed by Adequate Sleep: Participants were randomized to restrict sleep in phase 1 and crossed over to follow their habitual adequate sleep in phase 2
Period: Overall Study
Arm/Group | Adequate Sleep Followed by Sleep Restriction | Sleep Restriction Followed by Adequate Sleep
Started | 22 | 23
Completed | 16 | 20
Not Completed | 6 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adequate Sleep Followed by Sleep Restriction | Sleep Restriction Followed by Adequate Sleep | Total
Number analyzed (Participants) | 22 | 23 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.5 (12.3) | 31.6 (11.4) | 32.0 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 13 | 22
  Male | 13 | 10 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 16 | 22
  Not Hispanic or Latino | 16 | 7 | 23
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 7 | 9
  White | 13 | 8 | 21
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 2 | 5 | 7
Region of Enrollment [Number; unit: participants]
  United States | 22 | 23 | 45
Body fat volume by MRI [Mean (Standard Deviation); unit: Liter] — Population: MRI data were not obtained in one participant at baseline of phase 1 for sleep restriction
  Liter
    number analyzed (Participants) | 22 | 22 | 44
    (all) | 23.9 (10.1) | 24.6 (11.4) | 24.3 (10.7)
Sedentary Behavior [Mean (Standard Deviation); unit: minutes/day] | 741 (94) | 752.4 (93.4) | 746.4 (93.8)
Physical Activity [Mean (Standard Deviation); unit: minutes/day] — Population: Data were not available for 5 participants.
  minutes/day
    number analyzed (Participants) | 20 | 20 | 40
    (all) | 103.6 (49.5) | 89.3 (41.7) | 96.7 (46.5)
Ghrelin [Mean (Standard Deviation); unit: pg/mL] — Population: Blood samples were not available at baseline for 1 participant who started phase 1 in adequate sleep condition and 2 participants who started phase 1 in sleep restriction condition
  pg/mL
    number analyzed (Participants) | 21 | 21 | 42
    (all) | 870.3 (341.5) | 750.5 (251) | 810.4 (302.1)
Leptin [Mean (Standard Deviation); unit: ng/mL] — Population: Blood samples were not available at baseline for 1 participant who started phase 1 in adequate sleep condition and 1 participant who started phase 1 in sleep restriction condition
  ng/mL
    number analyzed (Participants) | 21 | 22 | 43
    (all) | 21.9 (19.3) | 26.5 (19.9) | 24.3 (19.5)
Glucagon-like peptide 1 [Mean (Standard Deviation); unit: pM] — Population: Blood samples were not available at baseline for 1 participant who started phase 1 in adequate sleep condition and 1 participant who started phase 1 in sleep restriction condition
  pM
    number analyzed (Participants) | 21 | 22 | 43
    (all) | 25.0 (13.1) | 21.5 (11.0) | 23.2 (12.1)
Orexin [Mean (Standard Deviation); unit: ng/mL] — Population: Assay was run on a sub-set of participants
  ng/mL
    number analyzed (Participants) | 15 | 17 | 32
    (all) | 1.34 (0.52) | 1.21 (0.48) | 1.28 (0.5)
Neuropeptide Y [Mean (Standard Deviation); unit: ng/mL] — Population: Assay was run on a subset of participants
  ng/mL
    number analyzed (Participants) | 15 | 17 | 32
    (all) | 1.37 (0.68) | 1.32 (0.68) | 1.34 (0.67)

OUTCOME MEASURES:

1. Primary Outcome: Endpoint Fat Volume
Description: Body composition (specifically fat volume) will be measured by MRI at baseline and endpoint.
Time Frame: Week 6 (endpoint)
Population: Data were available from 38 women who underwent MRI scanning for body composition assessment.
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Habitual Sleep (HS) | Sleep Restriction (SR)
Number analyzed (Participants) | 38 | 38
Liter | 24.0 (11.4) | 24.2 (11.6)

2. Secondary Outcome: Energy Expenditure (EE)
Description: EE is the amount of energy (or calories) that a person needs to carry out physical functions and will be assessed using Doubly Labeled Water (DLW), during the last 2 weeks of each sleep phase.
Time Frame: Measured over 14 days at the end of each phase (weeks 5 and 6; endpoint)
Measure: Mean (Standard Deviation); unit: kcal/d
Arm/Group | Habitual Sleep (HS) | Sleep Restriction (SR)
Number analyzed (Participants) | 32 | 30
kcal/d | 2445 (548) | 2476 (527)

3. Secondary Outcome: Physical Activity
Description: Time spent in moderate-to-vigorous physical activity.
Time Frame: Average over 6 weeks (measured daily)
Measure: Mean (Standard Deviation); unit: minutes/day
Arm/Group | Habitual Sleep (HS) | Sleep Restriction (SR)
Number analyzed (Participants) | 39 | 39
minutes/day | 86.1 (48.1) | 87.4 (43.4)

4. Secondary Outcome: Ghrelin
Description: Average post-baseline values
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Habitual Sleep (HS) | Sleep Restriction (SR)
Number analyzed (Participants) | 41 | 37
pg/mL | 856.6 (325.7) | 819.4 (287.2)

5. Secondary Outcome: Regional Brain Activation in Response to Food Stimuli
Description: The primary aim of this outcome was to investigate brain activation in response to food stimuli after a six-week period of Adequate Sleep (AS) or mild Sleep Restriction (SR). To achieve this, the investigators contrasted neuronal responses to food and non-food stimuli at two time points (baseline and six weeks post-intervention/control). This contrast allowed the investigators to calculate the number of voxels activated during the view of food stimuli compared to the number of voxels activated during the view of non-food stimuli (food - non-food) under each condition (AS or SR).
  Regional brain activation is reported as the total number of voxels activated on the group contrast images (combination of all analyzed participants) of the neuronal response to food stimuli compared to non-food stimuli. For this analysis, voxels were considered activated if they survived Gaussian Random Field theory correction with a 2-tailed p < 0.001 threshold when creating the group contrast images.
Time Frame: Week 6
Population: fMRI data was collected from 26 participants.
Measure: Number; unit: Activated Voxels
Groups:
- Participants Under Mild SR Conditions: Participants were randomized to a six-week period of adequate sleep.
- Participants Under AS Conditions: Participants were randomized to a six-week period of mild sleep restriction.
Arm/Group | Participants Under Mild SR Conditions | Participants Under AS Conditions
Number analyzed (Participants) | 26 | 26
Activated Voxels | 469 | 218

6. Secondary Outcome: Sedentary Behavior
Description: Time spent in sedentary physical activity.
Time Frame: Average over 6 weeks (measured daily)
Measure: Mean (Standard Deviation); unit: minutes/day
Arm/Group | Habitual Sleep (HS) | Sleep Restriction (SR)
Number analyzed (Participants) | 39 | 39
minutes/day | 766.9 (106.5) | 851 (87.6)

7. Secondary Outcome: Leptin
Description: Average post-baseline values
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Habitual Sleep (HS) | Sleep Restriction (SR)
Number analyzed (Participants) | 41 | 37
ng/mL | 23.4 (18.9) | 23.5 (19.2)

8. Secondary Outcome: Glucagon-like Peptide 1
Description: Average post-baseline values
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: pM
Arm/Group | Habitual Sleep (HS) | Sleep Restriction (SR)
Number analyzed (Participants) | 42 | 37
pM | 22.9 (9.7) | 23.0 (11.1)

9. Secondary Outcome: Orexin
Description: Average post-baseline values
Time Frame: 6 weeks
Population: Assays were run on a sub-set of participants.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Habitual Sleep (HS) | Sleep Restriction (SR)
Number analyzed (Participants) | 30 | 30
ng/mL | 1.29 (0.61) | 1.34 (0.62)

10. Secondary Outcome: Neuropeptide Y
Description: Average post-baseline values
Time Frame: 6 weeks
Population: Assay run on a sub-set of participants
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Habitual Sleep (HS) | Sleep Restriction (SR)
Number analyzed (Participants) | 29 | 29
ng/mL | 1.36 (0.70) | 1.41 (0.67)

11. Other Pre Specified Outcome: NIH Toolbox®
Description: Working memory data were collected using the List Sorting Working Memory Test from the NIH Toolbox. Data were transformed into a t-score ranging from 0-100 where a higher t-score indicates better performance. T-score of 50 indicates the population mean with a standard deviation of 10. Data were collected at baseline and after 6 weeks on study intervention. Traditionally, a clinically relevant threshold for cognitive data is 1.5 standard deviations below the mean. For a t-score, this would mean that a score of 35 or lower suggests clinical relevance.
Time Frame: Week 6 (endpoint)
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Habitual Sleep (HS) | Sleep Restriction (SR)
Number analyzed (Participants) | 12 | 10
T-score | 57.2 (6.5) | 50.8 (7.9)

12. Other Pre Specified Outcome: Neuro-behavioral Measures
Description: Episodic verbal learning and memory were collected using the Modified Rey Auditory Verbal Learning Test (ModRey). The primary variable of interest for this test is the number of correctly recalled words across three learning trials from List A consisting of 20 words in each trial. The total score range across three trials is 0-60. A higher score indicates better performance.
Time Frame: Week 6 (endpoint)
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Habitual Sleep (HS) | Sleep Restriction (SR)
Number analyzed (Participants) | 15 | 13
score | 33.8 (8.7) | 33.5 (9.5)

13. Other Pre Specified Outcome: Immune Function
Description: CD8+ T-cells from samples collected late in the day (non-fasted)
Time Frame: Week 5 (endpoint)
Measure: Mean (Standard Deviation); unit: cells/mL
Arm/Group | Habitual Sleep (HS) | Sleep Restriction (SR)
Number analyzed (Participants) | 11 | 13
cells/mL | 102212 (88785) | 107844 (259554)

14. Other Pre Specified Outcome: Immune Markers
Description: Classical monocytes measured from samples collected late in the day (non-fasted)
Time Frame: Week 5 (endpoint)
Measure: Mean (Standard Deviation); unit: cells/mL
Arm/Group | Habitual Sleep (HS) | Sleep Restriction (SR)
Number analyzed (Participants) | 11 | 13
cells/mL | 80038 (41470) | 134056 (59315)

15. Other Pre Specified Outcome: Distance Walked
Description: Distance walked over a 6-minute walk test
Time Frame: Week 5
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Habitual Sleep (HS) | Sleep Restriction (SR)
Number analyzed (Participants) | 28 | 29
meters | 620.2 (81.1) | 625.7 (85.2)

ADVERSE EVENTS:
Time Frame: Throughout participation in the study (from time accrued to end of phase 2); approximately 16-20 weeks for most participants.
Arm/Group | Habitual Sleep (HS) | Sleep Restriction (SR)
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/39
Other Adverse Events (participants affected / at risk) | 0/42 | 0/39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-05): https://cdn.clinicaltrials.gov/large-docs/76/NCT02960776/Prot_SAP_000.pdf